## Cover Page

Study Title: Homeless Youth Study - Stepping Stone Project

Document Type: Study Protocol with Statistical Analysis Plan (SAP)

Document Date: 6/24/18

## **Study Protocol**

The study will take 1 month and will consist of the following:

- Participants will complete a 1.5 hour enrollment session including the informed consent process, self-report questionnaires, phone set-up, and a phone usage and safety briefing.
- Over the course of 1 month, participants will have the opportunity to complete three 30-minute skills-based phone sessions with a Coach.
- Over the course of 1 month, participants will be asked to complete a daily survey and rate a daily tip via a mobile app.
- At the conclusion of the 1 month intervention, participants will complete another series of self-report questionnaires. If these questionnaires are completed, participants will receive another 5 months of paid phone service.

## **Statistical Analysis Plan**

- We will examine descriptive statistics of the number of contacts with the therapist, types of
  contact with the therapist, usage of the mobile applications, ratings of acceptability, ratings of
  perceived benefit, and ratings of interest in receiving mental health interventions via mobile
  technology.
- We will conduct paired t-tests to assess pre-post change in posttraumatic stress disorder, depression, anxiety, substance use, and risky behaviors.
- Algorithms will be developed in order to translate smartphone sensor data into meaningful outcomes. In particular, algorithms will be developed to evaluate the types of social communication that individuals use most often (e.g., talk, text, social media) and the extent to which communication serves a health-promoting (e.g., finding food) or health-diminishing function (e.g., acquisition of drugs).